CLINICAL TRIAL: NCT04972578
Title: Comparison of Gait in Syndesmosis Injuries Treated With Screw Fixation vs Suture Button
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Follow-up and consent was difficult and accrual was not being met.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0146-21-FB
Record Dates: First submitted 2021-04-23; First posted 2021-07-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Acute Disruption of Ankle Syndesmosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Screw Fixation (Active Comparator): Traditional fixation method of placing one or two screws across the syndesmosis.
  Interventions: Device: Suture Button vs Screw Fixation
- Suture Button (Active Comparator): Suture button implants which use a suture and anchor to repair the syndesmosis
  Interventions: Device: Suture Button vs Screw Fixation

INTERVENTIONS:
Device: Suture Button vs Screw Fixation — Syndesmotic fixation utilizing suture button fixation versus Screw Fixation (placing one or two screws across the syndesmosis)

SUMMARY:
Injuries to the distal tibiofibular syndesmosis are common and occur in an estimated 25% of all rotational ankle fractures. Anatomic reduction of the syndesmosis has been associated with improved functional outcome as well as decreased rates of posttraumatic arthritis. Both screw fixation and suture fixation have become accepted standards of care for treatment of syndesmotic injuries. Recent literature would suggest trends favoring suture fixation over screw fixation with improved quality of syndesmotic reduction, postoperative range of motion, and improved maintenance of syndesmotic reduction. However, the evidence remains heterogeneous, and patient reported outcomes have failed to show a superiority of one method over the other. Additionally, there have been no studies that demonstrate objective gait outcomes comparing screw versus suture fixation for syndesmotic injuries.

DETAILED DESCRIPTION:
This will be a prospective randomized study. Patients with isolated rotational ankle injuries with syndesmotic instability will be randomized to either screw fixation or suture fixation for treatment of their syndesmotic injury. Patients will be followed postoperatively for one year following surgery with documentation of both clinical outcomes and subjective patient reported outcomes. Additionally, postoperative gait patterns will be measured and compared between patients who had syndesmotic injuries treated with screw fixation versus suture fixation

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older
* Isolated rotational ankle injury
* Syndesmotic instability (determined either pre- or intra-operatively)
* Length-stable fibula fracture pattern

Exclusion Criteria:

* Open fracture
* Length-unstable fracture pattern (including Maisonneuve fracture pattern)
* Syndesmotic stability (determined either pre- or intra-operatively)
* Lower extremity neuropathy
* History of prior trauma or surgery to injured ankle
* Non-ambulatory
* Use of ambulatory assistive device prior to injury

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Gait parameter - Step length | 3 months
  Step length will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step length | 6 months
  Step length will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step length | 1 year
  Step length will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step width | 3 months
  Step width will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step width | 6 months
  Step width will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step width | 1 Year
  Step width will be measured in meters. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step time | 3 months
  Step time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step time | 6 months
  Step time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Step time | 1 year
  Step time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Swing time | 3 months
  Swing time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Swing time | 6 months
  Swing time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Swing time | 1 year
  Swing time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Stance time | 3 months
  Stance time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Stance time | 6 months
  Stance time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Stance time | 1 year
  Stance time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Double support time | 3 months
  Double support time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Double support time | 6 months
  Double support time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Double support time | 1 year
  Double support time will be measured in seconds. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Gait speed | 3 months
  Gait speed will be measured in meters per second. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Gait speed | 6 months
  Gait speed will be measured in meters per second. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.
Gait parameter - Gait speed | 1 year
  Gait speed will be measured in meters per second. Participants will walk down the length of a gait mat and back (20 feet in length, one-way). Five passes will be completed and the results averaged. Data will be collected on the Zeno Walkway using PKMAS software.

SECONDARY OUTCOMES:
Time to fracture union | 6 weeks, 3 months, 6 months, and 1 year
  Time to fracture union will be obtained based upon radiographic analysis at routine clinical follow-up visits.
Maintenance of syndesmotic reduction | 6 weeks, 3 months, 6 months, and 1 year
  Maintenance or loss of syndesmotic reduction will be evaluated radiographically at routine clinical follow-up visits.
Development of radiographic arthritis | 6 weeks, 3 months, 6 months, and 1 year
  Presence or absence of new radiographic tibiotalar arthritis will be noted on radiographs obtained at routine clinical follow-up visits.
Implant complications | 6 weeks, 3 months, 6 months, and 1 year
  Presence or absence of implant-related complications will be assessed radiographically at routine clinical follow-up visits (defined as screw fracture, loss of fixation, osteolysis surrounding implant).
Secondary procedures | 1 year
  The need for secondary procedures will be recorded. Secondary procedures would include of return trips to the OR for infection, for implant removal, for revision reduction or fixation, as well as in-office procedures including implant removal
Postoperative wound complications | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Presence or absence of wound complications will be evaluated on physical exam at routine clinical follow-up visits (defined as superficial or deep infection, delayed wound healing, wound dehiscence).
Ankle range of motion | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Ankle range of motion (tibiotalar dorsiflexion and plantarflexion) will be evaluated on physical exam at routine clinical follow-up visits (measured in degrees of dorsiflexion or plantarflexion from neutral).
Patient reported outcomes - PROMIS LE (Patient-Reported Outcomes Information System Lower Extremity) | 3 months, 6 months, and 1 year
  The PROMIS LE is a computer-adaptive test that reports a score of patient-perceived physical functioning (walking and mobility) specific to the lower extremity. Scores are reported as T scores, with a score of 50 equal to the mean of the general population. Higher scores indicate more favorable physical function. Theoretical maximum and minimum scores are 100 and 0, respectively.
Patient reported outcomes - Olerud-Molander Score | 3 months, 6 months, and 1 year
  The Olerud-Molander Score was designed to score patient-reported outcomes regarding symptoms after ankle fracture. Scale minimum and maximum are 0 and 100, respectively, with a higher score indicative of improved outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Putnam, MD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Nebraska Medicine, Bellevue Health Center, Bellevue, Nebraska
  - Lauritzen Outpatient Center, Omaha, Nebraska
  - Village Point Outpatient Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No